CLINICAL TRIAL: NCT01938911
Title: The Effects of Social Support and Oxytocin Administration on Physiological Stress Reactivity in Essential Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved away from Bern; lack of personnel in Bern to conduct the study within a reasonable time frame.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 215/10
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Essential Hypertension
Keywords: Trier social stress test; Oxytocin; Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Hypertensives with oxytocin and social support (Experimental): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Syntocinon-Spray; Behavioral: Social support
- Hypertensives with oxytocin without social support (Experimental): 80 normotensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Syntocinon-Spray
- Hypertensives without oxytocin with social support (Experimental): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Placebo of syntocinon; Behavioral: Social support
- Hypertensives without oxytocin or social support (Placebo Comparator): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Placebo of syntocinon
- Normotensives with oxytocin and social support (Experimental): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Syntocinon-Spray; Behavioral: Social support
- Normotensives with oxytocin without social support (Experimental): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Syntocinon-Spray
- Normotensives without oxytocin with social support (Experimental): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Placebo of syntocinon; Behavioral: Social support
- Normotensives without oxytocin or social support (Placebo Comparator): 80 hypertensive non-smoking medication-free men will be randomly assigned to receive intranasal OT (24 IU) or placebo 50 min before stress, and either social support (SS) from their best friend during the preparation period of the stress protocol or no social support.
  Interventions: Drug: Placebo of syntocinon

INTERVENTIONS:
Drug: Syntocinon-Spray — Intranasal oxytocin (24 IU)
  Arms: Hypertensives with oxytocin and social support; Hypertensives with oxytocin without social support; Normotensives with oxytocin and social support; Normotensives with oxytocin without social support
Drug: Placebo of syntocinon — Intranasal administration
  Arms: Hypertensives without oxytocin or social support; Hypertensives without oxytocin with social support; Normotensives without oxytocin or social support; Normotensives without oxytocin with social support
Behavioral: Social support — Social support from the best friend
  Arms: Hypertensives with oxytocin and social support; Hypertensives without oxytocin with social support; Normotensives with oxytocin and social support; Normotensives without oxytocin with social support

SUMMARY:
To test a psychopharmacological intervention strategy which may provide new insights into the mechanisms underlying the physiological hyperreactivity to stress observed in hypertension, we plan to test the effects of the neuropeptide oxytocin and social support on the neurobiological and psychological responsiveness to social stress. The study population for this project consists of 80 hypertensive and 80 normotensive non-smoking medication-free men. We expect exogenous oxytocin administration to enable hypertensives to effectively take advantage of the provided social support. Thereby, oxytocin may enhance the effect of social support on reducing the previously observed physiological hyperreactivity to stress in essential hypertensives.

DETAILED DESCRIPTION:
Background

Data on psychobiological stress reactivity in essential hypertension demonstrated physiological hyperreactivity to acute psychosocial stress in hypertensives as compared to normotensive controls in terms of sympathetic nervous system and hypothalamus-pituitary-adrenal axis activity, blood lipids, and coagulation activity. Moreover, we found lower perceived social support in hypertensives as compared to normotensives, with the highest physiological stress responses in hypertensives with low perceived social support.. In addition, the collaborating group of Prof. Heinrichs demonstrated that OT and social support interact to reduce neuroendocrine responses to stress in normotensive individuals. Given these findings and given the aforementioned hypothesized role for OT in physiological stress reactivity, particularly in hypertension, it seems promising to investigate the combined effects of OT and social support provision on physiological stress reactivity in essential hypertensives as compared to normotensives.

Objective

The proposed project will provide new information on neuroendocrine mechanisms underlying the observed physiological hyperreactivity to stress in essential hypertension. Moreover, stress reactivity of intermediate biological risk factors has not yet been investigated in experiments studying the effects of the acutely provided social support, either in healthy individuals or in hypertensives. The results of this project may provide important information for the development of effective interdisciplinary prevention and intervention strategies for essential hypertension

Methods

The methodological approach of social stress induction by the TSST used in our previous hypertension study will be translated to the planned project and we will repeatedly collect blood and saliva samples to measure neuroendocrine reactivity in terms of cortisol, epinephrine, and norepinephrine, as well as continuously measuring of heart rate and blood pressure. Blood pressure will be measured at each sampling timepoint as well as twice during the TSST (during the speech and during mental arithmetics). As our recent findings suggest strong associations between social support and heightened coagulation activity in healthy subjects before and after social stress, and as we found higher lipid and coagulation reactivity to psychosocial stress in hypertensives with catecholamine stress changes predicting elevated lipid stress reactivity, we plan to additionally measure biological risk factors for CHD.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years
* sufficient knowledge of German language in reading and understanding
* medication-free
* non-smoking
* systolic blood pressure ≥ 140 < 180 mmHg and/or diastolic blood pressure ≥ 90 < 110 mmHg for the hypertension group
* systolic blood pressure < 140 mmHg and diastolic blood pressure < 90 mmHg for the normotensive control
* written informed consent

Exclusion Criteria

* any alcohol, caffeine, and theine consumption 24 hours before the experiment
* regular strenuous exercise
* alcohol and illicit drug abuse
* liver and renal diseases
* chronic obstructive pulmonary disease
* allergies and atopic diathesis
* rheumatic diseases
* HIV
* cancer
* psychiatric and neurological diseases
* current infectious diseases

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in lipids from baseline | At 110 minutes

SECONDARY OUTCOMES:
Change in lipids from baseline | At 45, 80, 120, 130, and 170 minutes
Change in catecholamines from baseline | At 45, 80, 110, 120, 130, 140, 155, and 170 minutes
Change in cortisol from baseline | At 45, 80, 110, 120, 130, 140, 155, 170, 200, and 230 minutes
Change in cytokine level from baseline | At 45, 80, 110, 120, 200, and 230 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wirtz, Prof. Dr., Study Chair — University of Konstanz
Locations (1):
- Department of Psychology, University of Bern, Bern, Switzerland

REFERENCES:
- See also: Clinical Trial of effects of social support and oxytocin on physiological stress reactivity in essential hypertension — http://www.bioges.psy.unibe.ch/forschung/psychokardiologie/